CLINICAL TRIAL: NCT01521260
Title: Microbiological and Clinical Evaluation of Different Implant Surface Decontaminating Procedures in the Surgical Treatment of Peri-implantitis; a Double Blind Placebo Controlled Randomized Clinical Study
Brief Title: Implant Surface Decontamination in Peri-implantitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27147.042.09
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Peri-implantitis; Periodontal Disease
Keywords: dental implants; microbiology; chlorhexidine
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): Implants with peri-implantitis lesions will be surgically exposed, followed by a mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline, 1 minute of rinsing with a placebo solution (saline with appearance of chlorhexidine + CPC) and 1 minute of saline rinsing.
  Interventions: Procedure: placebo
- Chlorhexidine group (Active Comparator): Implants with peri-implantitis lesions will be surgically exposed, followed by a mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline, 1 minute of chemical cleansing using 0,12% chlorhexidine + cetylpyridinium chloride (CPC) without alcohol (Perio-aid®) and 1 minute of saline rinsing.
  Interventions: Procedure: Chlorhexidine

INTERVENTIONS:
Procedure: placebo — Implants with peri-implantitis lesions will be surgically exposed, followed by a mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline, 1 minute of rinsing with a placebo solution (saline with appearance of chlorhexidine + CPC) and 1 minute of saline rinsing.
  Arms: Placebo group
Procedure: Chlorhexidine — Implants with peri-implantitis lesions will be surgically exposed, followed by a mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline, 1 minute of chemical cleansing using 0,12% chlorhexidine + cetylpyridinium chloride (CPC) without alcohol (Perio-aid®) and 1 minute of saline rinsing.
  Other Names: Perio-aid
  Arms: Chlorhexidine group

SUMMARY:
Peri-implantitis is an infectious disease that resides in the mucosa surrounding dental implants and also affects the supporting bone. Because the number of implants placed in everyday clinical practice is continuously increasing, it is reasonable to anticipate an increasing prevalence of peri-implantitis. However, from the literature there is very little reliable evidence suggesting which could be the most effective interventions for treating peri-implantitis.

The primary objective of this controlled clinical study is to evaluate the microbiological effect of decontamination of the implant surface during the surgical treatment of peri-implantitis using a chlorhexidine or placebo solution. The secondary objectives are to assess both the clinical and the microbiological effectiveness of treatment of peri-implantitis.

It is hypothesized that rinsing of the implant surface using a 0.12% chlorhexidine solution does not lead to better microbiological and clinical results compared to rinsing with a placebo solution.

The present study is a double-blind, placebo-controlled, randomized clinical trial.

Adult patients with at least one endosseous implant in the oral cavity with clinical and radiographical signs of peri-implantitis will be included in this study.

Implants with peri-implantitis lesions will be surgically exposed, followed by mechanical cleansing using curettes and gauzes and cotton pellets soaked in saline followed by either 1 minute of rinsing with a placebo solution (saline with appearance of chlorhexidine) (control group) or 1 minute of chemical cleansing using 0,12% chlorhexidine + cetylpyridinium chloride (CPC) without alcohol (Perio-aid®) (test group). After 1 minute of saline rinsing the gingival flap will be returned slightly apical (in order to reduce pockets) and will be firmly sutured. For both groups the surgery is followed by 2 weeks of mouthrinses with 0,12% chlorhexidine + Cetylpyridinium Chloride (CPC) without alcohol (Perio-aid®) two times daily during 30 seconds.

The main study parameter is the microbial composition of the biofilm on the dental implant surface. Secondary study parameters are bleeding on probing, probing pocket depth, suppuration on probing, microbiological composition of the peri-implant sulcus, radiographic marginal bone level on standardized intraoral radiographs, presence of plaque, presence of calculus, marginal soft tissue recession implant failure, complications and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years of age
* The patient has at least one endosseous implant in the oral cavity with clinical and radiographical signs of peri-implantitis. Peri-implantitis is defined as a loss of marginal bone ≥ 2 mm as compared to a fixed reference point on the dental implant, in combination with bleeding and/or suppuration on probing and a peri-implant probing depth ≥ 5 mm;
* The implants have been exposed to the oral environment for at least two years;
* The patient is capable of understanding and giving informed consent.

Exclusion Criteria:

* Medical and general contraindications for the surgical procedures;
* A history of local radiotherapy to the head and neck region;
* Pregnancy and lactation;
* Diabetes;
* Systemic use of antibiotics during the last 3 months;
* Long-term use of anti-inflammatory drugs;
* Incapability of performing basal oral hygiene measures as a result of physical or mental disorders;
* Active, uncontrolled periodontal pathology of the remaining dentition;
* Local use of antibiotics or use of other anti-septic / antimicrobial therapies in the oral cavity during the last 3 months;
* Use of mouthrinses;
* Bruxism;
* Implants placed in skin grafted areas;
* Implants with bone loss due to other reasons than bacterial infection (e.g. loose screw, inadequate positioning of the implant);
* Implants with bone loss exceeding 2/3 of the length of the implant or implants with bone loss beyond the transverse openings in hollow implants;
* Implant mobility;
* Implants at which no position can be identified where proper probing measurements can be performed;
* Previous surgical treatment of the peri-implantitis lesions;
* Previous non-surgical treatment of the peri-implantitis lesions during the last 6 months (scaling or curretage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne CM de Waal, dds, Principal Investigator — University Medical Center Groningen; Arie Jan van Winkelhoff, prof. dr., Study Chair — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: october 2009-september 2010 location: University Medical Center Groningen
Pre-assignment Details: Assessed for eligibility:55 patients Excluded 25, because 'not meeting inclusion criteria (n=20) or 'declined to participate' (n=5)
Period: Overall Study
Arm/Group | Placebo Group | Chlorhexidine Group
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Chlorhexidine Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.0) | 59.4 (14.0) | 60.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Netherlands | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Bacterial Load on the Exposed Implant Surface
Description: Total bacterial load as obtained by sweeping a microbrush across the implant surface after flap deflection. Samples are obtained immediately after flap deflection and granulation tissue removal AND after the decontamination procedure (mechanical debridement, rinsing of the implant surface using the placebo or chlorhexidine solution, saline rinsing) but before flap closure. The log-transformed mean change in bacterial load is calculated (difference between the two time points --> difference in sample BEFORE decontamination and AFTER decontamination procedure).
Time Frame: During the surgical procedure: 1. immediately after flap deflection and granulation tissue removal AND 2. after the decontamination procedure but before flap closure.
Measure: Log Mean (Standard Deviation); unit: log (colony forming units/ml)
Units Other Than Participants: implants
Arm/Group | Placebo Group | Chlorhexidine Group
Number analyzed (Participants) | 15 | 15
Number analyzed (implants) | 35 | 25
log (colony forming units/ml) | 2.77 (2.12) | 4.21 (1.89)

2. Secondary Outcome: Bleeding on Probing
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

3. Secondary Outcome: Probing Pocket Depth
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

4. Secondary Outcome: Suppuration on Probing
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

5. Secondary Outcome: Microbiological Composition of the Peri-implant Sulcus
Time Frame: baseline (T0), 3 and 12 months after intervention (T3, T12)
Reporting Status: Not Posted

6. Secondary Outcome: Radiographic Marginal Bone Level on Standardized Intraoral Radiographs
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

7. Secondary Outcome: Presence of Plaque
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

8. Secondary Outcome: Presence of Calculus
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

9. Secondary Outcome: Marginal Soft Tissue Recession
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

10. Secondary Outcome: Implant Failure
Description: defined as implant mobility of previously clinically osseointegrated implants and removal of non-mobile implants because of progressive marginal bone loss or infection
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

11. Secondary Outcome: Complications and Adverse Events
Time Frame: baseline (T0), 3, 6 and 12 months after intervention (T3, T6, T12)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo Group | Chlorhexidine Group
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes